CLINICAL TRIAL: NCT06043076
Title: The Effect of Intermittent Theta-Burst Stimulation on Motor Cortical Plasticity, Blood Glucose, and Cardiovascular Response in Healthy Young Adults
Brief Title: iTBS Effect on M1 Plasticity, Blood Glucose, and Cardiovascular Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wan Aliaa Wan Sulaiman, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: JKEUPM-2023-674
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy Young Adults
Keywords: Transcranial magnetic stimulation (TMS); Intermittent theta-burst stimulation (iTBS); Primary motor cortex (M1); Neuroplasticity; Heart rate; Blood pressure; Blood glucose; Healthy; Young adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active then sham stimulation (Experimental): Active iTBS over the left M1 hand region, followed after 1 week washout period by sham iTBS over the left M1 hand region
  Interventions: Device: TMS; Device: Sham
- Sham then active stimulation (Experimental): Sham iTBS over the left M1 hand region, followed after 1 week washout period by active iTBS over the left M1 hand region
  Interventions: Device: TMS; Device: Sham

INTERVENTIONS:
Device: TMS — Active iTBS will be applied using a butterfly figure-of-eight C-B60 coil connected to MagPro R30 stimulator with add-on Theta Burst option (MagVenture A/S, Farum, Denmark).
Device: Sham — Sham iTBS will be applied using acoustic stimulation of a second coil behind the participant's head

SUMMARY:
Transcranial magnetic stimulation is a medical device that can alter motor cortical (M1) excitability through the scalp via various protocols. Among these, intermittent theta-burst stimulation (iTBS) is a novel protocol that enhances the M1 excitability for several minutes beyond stimulation. The changes in M1 excitability might in turn be accompanied by other physiological responses in the human body. This study will explore the effect of iTBS protocol on M1 plasticity, heart rate, blood pressure, and blood glucose in healthy young adults in comparison to sham stimulation.

ELIGIBILITY:
Inclusion criteria:

* Healthy young adults (18-35 years old)
* Right-handed
* Fully vaccinated against COVID-19

Exclusion criteria:

* Subjects with contraindications to TMS based on the screening 13-item questionnaire for TMS candidacy
* Smokers
* Obese (BMI ≥ 30)
* Highly active subjects
* Active or previous lab-confirmed COVID-19 with long symptoms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) | Pre-iTBS (baseline) and post-iTBS at 5,10,20, and 30 minutes
  Peak-to-peak MEP amplitude elicited by single-pulse TMS over the left M1 representation of the first dorsal interosseous (FDI) muscle. In each MEP measurement throughout the study, a total of 12 MEP readings, elicited by single pulse TMS at an intensity of 120% resting motor threshold, and separated by 15 seconds, will be collected.
  In each time point post-iTBS, the mean value of MEPs (aka, conditioned MEPs) will be averaged and compared to pre-iTBS (aka, baseline MEPs) using the following equation:
  (conditioned MEP amplitude/baseline MEP amplitude) × 100. A value of 90-110% represents no change, while values < 90% represent suppression, and > 110% represent facilitation of the M1 plasticity following iTBS.

SECONDARY OUTCOMES:
TMSens_Q questionnaire | At the end of every session
  Self-reported side effects using structured TMSens_Q questionnaire to evaluate the tolerability of iTBS
Blood glucose | Pre-iTBS (baseline) and post-iTBS at 0 and 30 minutes
  Capillary blood glucose using portable glucometer
Blood pressure | Pre-iTBS (baseline) and post-iTBS at 0 and 30 minutes
  Systolic blood pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Pressure (MAP) using semi-automated oscillometric sphygmomanometer. Unit of measure: mmHg
Heart rate | Pre-iTBS (baseline) and post-iTBS at 0 and 30 minutes
  Heart rate (bpm) using semi-automated oscillometric sphygmomanometer
Baseline corticospinal excitability indices | Baseline
  Test-retest reliability of resting motor threshold (RMT) and MEP amplitude

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw datasets collected during the trial will be freely available upon completion on the Open Science Framework repository at https://osf.io/
URL: https://osf.io/